CLINICAL TRIAL: NCT03797300
Title: Accuracy of Pulse Oximeters With Profound Hypoxia
Brief Title: Pulse Oximeter and Respiratory Rate Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spry Health (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SpryUCSF2
Record Dates: First submitted 2019-01-02; First posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Hypoxia; Hypercapnia; Hypocapnia
MeSH Terms: conditions — Hypoxia; Hypercapnia; Hypocapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Primary (Experimental)
  Interventions: Device: Spry Loop Band

INTERVENTIONS:
Device: Spry Loop Band — Loop band measures pulse oximetry and respiration rate

SUMMARY:
Assessment of Spry Health's Loop oximetry accuracy in profound hypoxia Assessment of Spry Health's Respiratory rate accuracy in normal conditions and profound hypoxia

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult willing to participate

Exclusion Criteria:

* Wrist size outside the indicated use
* Low perfusion
* Smoking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Accuracy of SpO2 measurement | duration of subject monitoring, usually up to one hour
  Pulse oximetry measurement accuracy vs. gold standard
Accuracy of Respiratory Rate measurement | duration of subject monitoring, usually up to one hour
  Respiratory rate measurement accuracy vs. gold standard

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Hypoxia Lab, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No